CLINICAL TRIAL: NCT04740385
Title: Role of Transthoracic Lung Ultrasound in Confirmation of Correct Double Lumen Endotracheal Tube
Brief Title: Role of Lung Ultrasound in Confirmation of Correct Double Lumen Endotracheal Tube Placement in Thoracic Surgeries
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Other Study IDs: 202101-2P-02002
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Diagnostic Accuracy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients: Correct position of double lumen endotracheal tube will be assessed using lung sonography, routine chest auscultation and fiberoptic brochoscopy
  Interventions: Diagnostic Test: Lung auscultation; Device: Fiberoptic bronchoscopy; Device: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung auscultation — auscultation of air entry through chest wal
Device: Fiberoptic bronchoscopy — Checking correct double lumen position through direct vision using fiberoptic bronchoscopy
Device: Lung Ultrasound — real time visualization of air entry to the lungs using trans-thoracic lung ultrasound

SUMMARY:
to assess the efficacy of lung ultrasound versus conventional auscultation method and fiberoptic bronchoscopy in confirmation of double lumen tube position

DETAILED DESCRIPTION:
Confirmation of double lumen tube position by auscultation followed fiberoptic bronchoscopy then lung ultrasound. After double lumen intubation all patient tube position will be confirmed using auscultation then fiberoptic bronchoscopy then lung ultrasound

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgeries under general anesthesia requiring double lumen endotracheal intubation
* ASA I-II

Exclusion Criteria:

* patient refusal
* patients not meeting the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer patients undergoing thoracic surgeries requiring double lumen intubation
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of lung ultrasound in confirmation of correct double lumen position | 5 minutes
  real time visulaization of air entry to the lung

SECONDARY OUTCOMES:
procedural time | 5 minutes
  time taken to confirm tube position

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer
Locations (1):
- Department of anesthesia and pain medicine. National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided